CLINICAL TRIAL: NCT06289140
Title: Evaluation of the Oral Bioavailability of a New Formulation of Pterostilbene Co-crystal in Comparison With Its Free Form in Healthy Volunteers: Crossover, Randomized and Simple Blind Study (BIOPTERO2)
Brief Title: Oral Bioavailability of a New Formulation of Pterostilbene Cocrystal in Comparison With Its Free Form (BIOPTERO2)
Acronym: BIOPTERO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: Circe, S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BIOPTERO2
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Biological Availability
Keywords: Polyphenols; Antioxidant activity; Co-crystallization; Pterostilbene; Oral bioavailability
MeSH Terms: interventions — Gelatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pterostilbene cocrystal - gelatin capsule (Experimental): Participants consuming one gelatin capsule of Pterostilbene cocrystal (ccPT)
  Interventions: Dietary Supplement: Pterostilbene cocrystal (ccPT) - Gelatin capsule
- Pterostilbene cocrystal - gastro-resistant capsule (Experimental): Participants consuming one gastro-resistant capsule of Pterostilbene cocrystal (ccPT)
  Interventions: Dietary Supplement: Pterostilbene cocrystal (ccPT) - Gastro-resistant capsule
- Pterostilbene free form (Active Comparator): Participants consuming one capsule with Pterostilbene free form (PT)
  Interventions: Dietary Supplement: Pterostilbene free form (PT)

INTERVENTIONS:
Dietary Supplement: Pterostilbene cocrystal (ccPT) - Gelatin capsule — Participants will intake one gelatin capsule with 75 mg of Pterostilbene cocrystal (ccPT).
  Arms: Pterostilbene cocrystal - gelatin capsule
Dietary Supplement: Pterostilbene free form (PT) — Participants will intake one capsule with 50 mg of Pterostilbene free form (PT)
  Arms: Pterostilbene free form
Dietary Supplement: Pterostilbene cocrystal (ccPT) - Gastro-resistant capsule — Participants will intake one gastro-resistant capsule with 75 mg of Pterostilbene cocrystal (ccPT).
  Arms: Pterostilbene cocrystal - gastro-resistant capsule

SUMMARY:
The goal of this interventional study is to to evaluate the oral bioavailability of the crystallized form of pterostilbene (ccPT) compared to its commercial free base form (pterostilbene (PT) in healthy volunteers. The main question it aims to answer are:

• Do the crystallized forms of pterostilbene (ccPT) using two different encapsulation methods exhibit greater bioavailability than its commercial free base form (PT)?

Participants will attend to four visits: a preselection visit (V0), a visit for the first postprandial study (V1), a visit for the second postprandial study (V2) after one-week washing period and a visit for the third postprandial study (V3) after another one week washing period.

Researchers will analyze the three postprandial assays to determine which type of ccPT encapsulation provides the highest bioavailability compared to the commercial free base form (PT).

DETAILED DESCRIPTION:
The oxidative stress (OS) is a condition where pro-oxidative processes overwhelm cellular antioxidant defenses due to disruption in redox signaling. This results in the body's inability to eliminate reactive oxygen species (ROS) or repair damages, potentially leading to severe impacts on cells, tissues, and organs.

Pterostilbene (PT) is a stilbenoid found in various natural sources, emerging as an antioxidant with potential preventive and therapeutic properties in numerous diseases. Despite its promising properties, PT's low water solubility and bioavailability pose challenges.

Nutraceutical co-crystallization is a recent strategy to enhance solubility and oral bioavailability. It has been identified that a new pterostilbene:picolinic acid (1:1) co-crystal, significantly increasing solubility and oral bioavailability compared to commercial free base PT.

The study aims to evaluate oral bioavailability (AUC0-24h) of PT (free and total) from ccPT compared to commercial PT, using two different encapsulation methods. Secondary objectives include determining pharmacokinetic parameters such as AUCinf, relative oral bioavailability (Frel), Cmax, Tmax, and T1/2 for both free and total PT.

This randomized, crossover, single-blind clinical trial aims to provide insights into the effectiveness of the new ccPT formulation in enhancing PT's oral bioavailability compared to the commercial PT formulation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 65 years of age.
* Sign the informed consent form.
* Know how to read, write and speak Spanish

Exclusion Criteria:

* Take supplements or multivitamin supplements or phytotherapeutic products (especially infusions) that interfere with the treatment under study up to 30 days before the start of the study.
* Be lacto-vegetarian, lacto-ovo-vegetarian, or vegan.
* Present intolerances and/or food allergies related to pterostilbene or the excipients.
* Be a smoker.
* Having received antibiotic treatment up to 30 days before the start of the study.
* Present values of body mass index ≤ 18kg/m^2 or ≥ 35 kg/m^2.
* Present some chronic disease with clinical manifestations: coronary heart disease, cardiovascular disease, diabetes, celiac disease, Crohn's disease, chronic kidney disease, cancer, autoimmune diseases (such as fibromyalgia), respiratory and/or gastrointestinal diseases that may compromise the absorption of the compound.
* Clinical history of anemia.
* Being pregnant or intending to became pregnant.
* Be in breastfeeding period.
* Being unable to follow the study guidelines.
* Participate in or have participated in a clinical trial or nutritional intervention study in the last 30 days before inclusion in the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Bioavailability of Pterostilbene calculated by area under the curve (AUC 0-24) of plasma pterostilbene levels, both free and total. | At week 1, week 2 and week 3
  Fasting pterostilbene levels in plasma will be determined by liquid chromatography coupled to mass spectrophotometry before consume the capsule with pterostilbene until 24 hours postprandially at 8 points after consuming the capsule (0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours and 24 hours).
  Total PT will be quantified indirectly after hydrolysis of the conjugated glucuronide and sulfate metabolites to free PT in the presence of β-glucuronidase and arylsulfatase in the plasma samples.

SECONDARY OUTCOMES:
Area under the curve (AUC 0-inf) of plasma pterostilbene levels, both free and total. | At week 1, week 2 and week 3
  Fasting pterostilbene levels in plasma will be determined by liquid chromatography coupled to mass spectrophotometry before consume the capsule with pterostilbene until 24 hours postprandially at 8 points after consuming the capsule (0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours and 24 hours).
  Total PT will be quantified indirectly after hydrolysis of the conjugated glucuronide and sulfate metabolites to free PT in the presence of β-glucuronidase and arylsulfatase in the plasma samples.
Relative bioavailability of plasma pterostilbene levels (Frel). | At week 1, week 2 and week 3
  Relative bioavailability of plasma pterostilbene levels, both free and total
Maximum plasma concentration (Cmax) | At week 1, week 2 and week 3
  Maximum plasma concentration of pterostilbene, total and free.
Time for maximum plasma concentration (Tmax) | At week 1, week 2 and week 3
  Time period for the maximum plasma concentration of pterostilbene, both total and free.
Half-life (T1/2). | At week 1, week 2 and week 3
  Time taken for half the initial dose of pterostilbene, both total and free, administered to be eliminated from the body.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari, PhD, Principal Investigator — Fundació Eurecat
Locations (1):
- Fundació Eurecat, Reus, Spain

IPD SHARING:
Plan to Share IPD: No
In this study IPD will not be shared with other researchers because all the information will be processed by the UTNS of Eurecat.

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org